CLINICAL TRIAL: NCT04782466
Title: Physical Activity, Quality of Life and Disease Outcomes in Youth With Multiple Sclerosis: the ATOMIC (Active Teens Multiple Sclerosis) Physical Activity Research Program
Brief Title: ATOMIC (Active Teens Multiple Sclerosis) Physical Activity Research Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Alabama at Birmingham (Other); Queen's University (Other); National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, E. Ann Yeh, Senior Associate Scientist, Division of Neuroscience and Mental Health, SickKids Research Institute, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1000065261; RG-1901-33188 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-05

CONDITIONS: Pediatric Multiple Sclerosis
Keywords: Physical Activity; Exercise; Multiple Sclerosis; Demyelinating Disorders; Pediatric; Neurology; Children
MeSH Terms: conditions — Motor Activity; Multiple Sclerosis; Demyelinating Diseases | interventions — Exercise; Methods

STUDY DESIGN:
Intervention Model Description: At baseline, participants will be randomized using online research randomizer software, in blocks of 2 each, balanced for the clinical site, sex, and pubertal status (using self-selected Tanner staging), which may independently predict physical fitness level and has also been associated with physical activity level especially in adolescent girls to either a 6-month PA intervention or waitlist attention-control condition. The research coordinator will request the randomization of the participant as provided by the online research randomizer at the completion of the baseline test and will inform the study participant of their assigned study arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will receive both the intervention and the attention-control condition and will not be informed of which of the procedures is the active intervention condition. The statistician, PI, and fitness testers, and physical activity data analysts will be blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The participant receives the intervention immediately following baseline measurements.
  Interventions: Behavioral: Physical Activity (PA) Intervention
- Waitlist attention-control (Other): The participant receives the control condition for 6 months following baseline measurements. After 6 months, the baseline measurements are repeated and then the participant receives the intervention.
  Interventions: Behavioral: Waitlist attention-control

INTERVENTIONS:
Behavioral: Physical Activity (PA) Intervention — The ATOMIC intervention consists of four primary components: one-on-one chats with a PA coach, informational posts, PA self-monitoring through an activity tracker and educational modules regarding different aspects of becoming PA delivered through the MS-specific PA app. An overarching goal of moving youth with MS towards meeting current Moderate to Vigorous Physical Activity (MVPA) recommendations will be used in addition to initial results from accelerometer monitoring and evaluation of current PA intentions to establish step goals, with planned weekly incremental increases (10% weekly to goal).
  Arms: Intervention
Behavioral: Waitlist attention-control — For a period of 6-months, participants will receive the control conditions that involve contact from study personnel and a nutritional educational module to ensure equivalent social contact in both arms of the study. After the 6-months, participants will receive the same intervention as the intervention arm.
  Arms: Waitlist attention-control

SUMMARY:
The investigators have previously shown that youth with MS are very inactive, and that vigorous physical activity is associated with higher levels of well-being and lower MS disease activity in youth. Yet, no effective physical activity interventions have been developed for youth with MS to date. The investigators have taken input from youth with MS to create a Smartphone-based app (the ATOMIC - Active Teens with Multiple Sclerosis - App) that provides tailored physical activity information and coaching, provides tools to increase social connectedness, and promotes physical activity. This proposed research will therefore address the problem of inactivity in youth with MS by studying an intervention to increase physical activity.

DETAILED DESCRIPTION:
Youth with MS have highly active disease and report high levels of fatigue and depression. As MS is a lifetime diagnosis, amelioration of these outcomes may have a sustained and important effect on the lives of these youth. Effective interventions oriented towards improving these outcomes are therefore imperative to develop and study. Importantly, recent work suggests that increased PA has the potential to improve brain tissue integrity, re-myelination, mental health outcomes, and quality of life in youth with MS. The investigators have demonstrated associations between lower levels of PA and higher levels of depressive symptoms and fatigue in these youth over time. Furthermore, the investigators have demonstrated an association between higher levels of PA and lower levels of disease activity in youth with MS. Importantly, preliminary work by the investigators shows that youth with MS have very low levels of PA. Increasing PA, therefore, has the potential to have both disease-modifying and psychosocial benefits in youth with MS.

The investigators have developed a user-driven app and program, the ATOMIC intervention, which addresses barriers to PA participation the investigators previously identified. The program provides youth with tools to increase goal setting, PA self-efficacy, and knowledge, and is embedded in a youth-focused app that is supported by health coaches. Notably, in preliminary work, the investigators have found the ATOMIC program to be acceptable to youth, and furthermore, that it was associated with a 31% increase in physical activity.

These strong preliminary results support moving forward with this proposed research, a multi-center randomized wait-list controlled trial (RCT) of the ATOMIC mobile app and coaching-based physical activity (PA) intervention in youth with multiple sclerosis (MS). The proposed study will examine the extent to which the intervention can change PA levels in this cohort. Additional goals will be to evaluate the effect of the ATOMIC intervention on behavioural change mediators, fitness, and psychosocial outcomes.

For this study, the investigators will recruit 56 youth with MS followed at three tertiary children's hospitals with large, established pediatric MS programs: The Hospital for Sick Children, Children's Hospital of Philadelphia, and the University of Alabama at Birmingham.

ELIGIBILITY:
Inclusion Criteria:

1. Youth 11-21 years of age;
2. MS diagnosis or clinically isolated syndrome, as per revised McDonald diagnostic criteria and International Pediatric MS Study Group criteria prior to the age of 18;
3. Participating in less than three hours of structured physical activity per week.

Exclusion Criteria:

1. Have non-specific white matter abnormalities and metabolic or infectious etiologies for white matter abnormalities;
2. Do not speak and read English at a level needed to complete the questionnaires (4th grade level);
3. Have significant motor disability, classified as an Expanded Disability Status Scale (EDSS) ≥4;
4. Are at increased risk of cardiac or other complications of exercise testing (e.g. cardiac disease, diabetes), as determined by the pediatric neurologist or physician.

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Level | Entire study - up to 18 months
  Accelerometry is a valid device-based physical activity measurement tool that will be used to determine physical activity. Children will be asked to wear the accelerometer daily for a week, and the investigators will analyze cases that have four or more days of data with ≥10 hours of wear time per day. The investigators will process the accelerometer data and use step counts as well as validated cut-offs to determine time spent in sedentary, light, and Moderate to Vigorous Physical Activity (MVPA) (minutes/day). The focus of the investigators will be to determine the effect of the ATOMIC intervention on device-measured physical activity levels.

SECONDARY OUTCOMES:
Aerobic Capacity | Entire study - up to 18 months
  The investigators will determine cardiorespiratory fitness by measuring peak oxygen uptake (VO2Peak) using a maximal exercise test on a cycle ergometer.
Self-Reported PA Outcomes | Entire study - up to 18 months
  The Godin Leisure-Time Exercise Questionnaire (GLTEQ) will be used to self-report physical activity outcomes. This self-report 7-day activity recall scale has been validated in the pediatric population and in the pediatric MS population.
Social Cognitive Theory Based Mediators of Physical Activity | Entire study - up to 18 months
  This is a composite set of questionnaires used to evaluate Social Cognitive Theory (SCT) based mediator. The focus of the investigators will be to determine the effect of the intervention on social cognitive theory mediators of PA.

OTHER OUTCOMES:
Tertiary Outcome Measures: Depression | Entire study - up to 18 months
  The Centre for Epidemiological Studies Depression Scale Children's Rating Scale (CES-DC) is a valid and reliable 20-item, self-rated, symptom-oriented scale suitable for people aged six to 23.
Tertiary Outcome Measures: Quality of Life | Entire study - up to 18 months
  The Varni Pediatric Quality of Life Inventory - Core Module (PedsQL) is a 23-item scale that measures social, physical, emotional, school functioning quality of life that has been shown to be a valid and reliable measure of quality of life in children with chronic conditions.
Tertiary Outcome Measures: Fatigue | Entire study - up to 18 months
  The Varni Pediatric Multidimensional Fatigue Scale (PedsQL-MFS) is a validated and reliable 18-item, self-rated (parent and self-report), symptom-oriented scale suitable for youths aged 8 to 18 that includes fatigue subscales (general, sleep/rest and cognitive fatigue).
Tertiary Outcome Measures: Cognitive Function | Entire study - up to 18 months
  The Symbol Digit Modalities Test (SDMT) is a widely used, validated paper and pencil neurocognitive test which assesses processing speed (i.e. the speed of thinking). It validated and used widely in pediatric multiple sclerosis.
Tertiary Outcome Measures: Anxiety | Entire study - up to 18 months
  The Screen for Anxiety Related Disorders (SCARED) scale is a validated and reliable 41-item, self-rated, symptom score suitable for youths ages 9 to 18.

CONTACTS AND LOCATIONS:
Overall Officials: E. Ann Yeh, MA, MD, FRCPC, Dip ABPN, Principal Investigator — The Hospital for Sick Children
Locations (3):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuroinflammatory Disorders Program Research Website — https://lab.research.sickkids.ca/neuroinflamm/